CLINICAL TRIAL: NCT01192971
Title: Randomized, Open-label, Multi-center, Phase II Study of Apatinib in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of Apatinib in Patients With Advanced Hepatocellular Carcinoma
Acronym: HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Eighty-One Hospital of People's Liberation Army (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HENGRUI20100510
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: HCC, Apatinib, phase II, Cancer
MeSH Terms: conditions — Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: 850mg (Experimental): A: Experimental apatinib 850 mg qd p.o, and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Apatinib
- B: 750mg (Experimental): B: Apatinib 750 qd p.o. and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — apatinib p.o. once daily for 4 weeks

SUMMARY:
This phase II trial will be studying how well Apatinib working in patients with Hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologic confirmed advanced hepatocellular carcinoma
* Patients who are unable to or unwilling to undergo surgery or interventional procedures via hepatic artery, or patients who have relapsed/progressed after surgery or interventional procedure via hepatic artery for ≥ 4 weeks and are unable to use sorafenib.
* Life expectancy of more than 12 weeks.
* ECOG performance scale 0 - 2.
* Child -Pugh score A，BCLC stage B or C.
* At least one therapy naïve measurable lesion (larger than 10 mm in diameter by spiral CT scan, conforming to RECIST 1.1).
* Have not received systemic chemotherapy or molecular targeted therapy. At least 4 weeks must have elapsed for patients who have previously underwent radiotherapy or surgery, and all the adverse drug reactions (ADRs) or wounds have completely healed. At least 6 months must have elapsed for patients who have received adjuvant chemotherapy.
* Adequate organ functions (hemoglobin≥ 90g/L ,platelets ≥80 × 109/L, neutrophil≥ 1.5 × 109/L, albumin ≥ 29 g/L, Plasma creatinine ≤ 1.5 × ULN , ALT and AST< 5 × ULN; TBIL ≤ 1.5 × ULN.
* Signed and dated informed consent.Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with known intrahepatic cholangiocarcinoma, mixed hepatocellular carcinoma, and fibrolamellar hepatocellular carcinoma; other malignancies previously or currently, except for cured skin basal cell carcinoma and cervical carcinoma in situ.
* Dysphagia, chronic diarrhea, and intestinal obstruction, which significantly affect drug intake and absorption.
* Evidence of CNS metastasis.
* Subjects with hypertension which cannot be well controlled by antihypertensives; grade II or greater myocardial ischemia or myocardial infarction, poorly controlled arrhythmia, and cardiac insufficiency grades III to IV according to NYHA criteria; cardiac color Doppler ultrasound examination: LVEF (left ventricular ejection fraction) of < 50%.
* Subjects with abnormal coagulation functions, and the tendency of bleeding or those who are currently treated by a thrombolytic or anticoagulant therapy.
* Definite concern of gastrointestinal hemorrhage, and history of gastrointestinal hemorrhage within 6 months.
* Patients with symptomatic ascites requiring therapeutic paracentesis or drainage, or with a Child-Pugh score of ≥ 2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
TTP (Time to Progression) | 8 weeks

SECONDARY OUTCOMES:
Overall Survival | 8 weeks
DCR (Disease control rate | 8 weeks
ORR (objective response rate) | 8 weeks
Serum alpha-fetoprotein (AFP) level | 8 weeks
QoL (quality of life): EORTC QLQ-C30 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shukui Qin, Dr, Principal Investigator — Nanjing Millitary Eighty-one Hosiptal
Locations (1):
- Nanjing Millitary Eighty-one Hosiptal, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided